CLINICAL TRIAL: NCT02248467
Title: Study of the Effect of Testosterone Replacement Therapy on Metabolic Parameters, Prostatic Inflammation Symptoms and Lower Urinary Tract Symptoms (LUTS) in Hypogonadal Obese Subjects Eligible for Bariatric Surgery.
Brief Title: Study of the Effect of Testosterone Treatment on Metabolic Parameters and Urinary Symptoms in Bariatric Patients
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, Full Professor of Endocrinology, University of Florence
Other Study IDs: ANDRO-AOUC-2013-01
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Hypogonadism; Prostatic Hyperplasia; Insulin Resistance
Keywords: Testosterone replacement therapy
MeSH Terms: conditions — Obesity; Hypogonadism; Prostatic Hyperplasia; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- eugonadal: 50 eugonadal subjects
- untreated hypogonadal: 25 asymptomatic hypogonadal subjects
- treated hypogonadal: 25 symptomatic hypogonadal subjects treated - In the present study, we decided to monitor only sexual symptoms of androgen deficiency due to the fact that testosterone replacement therapy (TRT) should be expected to improve them in the time span until surgery. These patients will be treated with TRT as per clinical practice.

SUMMARY:
The primary purpose of the study is to evaluate, in obese and hypogonadal patients eligible for bariatric surgery, the effect of testosterone replacement therapy in improving lower urinary tract symptoms (LUTS) assessed using the IPSS (International Prostate Symptom Score) questionnaire, compared to hypogonadal untreated subjects and eugonadal subjects.

DETAILED DESCRIPTION:
Primary objective:

- Evaluation in obese and hypogonadal patients candidates for bariatric surgery of the effect of testosterone replacement therapy in improving the symptoms of LUTS (assessed using the IPSS questionnaire) compared to hypogonadal untreated subjects and eugonadal subjects.

Secondary objectives:

* Evaluation of the effect of testosterone in obese and hypogonadal patients candidates for bariatric surgery in improving metabolic parameters (glycaemia, oral glucose tolerance test, HbA1c, total cholesterol, HDL cholesterol, triglycerides, arterial pressure, BMI, waist circumference) compared to hypogonadal untreated subjects and eugonadal subjects
* Evaluation of the effect of testosterone in obese and hypogonadal patients candidates for bariatric surgery in improving uroflowmetric parameters compared to hypogonadal untreated subjects and eugonadal subjects
* Evaluation of the effect of testosterone in obese and hypogonadal patients candidates for bariatric surgery on the ultrasound characteristics of the prostate (macro-calcifications, intraprostatic arterial velocity, volume of the prostate gland).
* Evaluation of the effect of testosterone in obese and hypogonadal patients candidates for bariatric surgery on pre-adipocytes isolated from visceral adipose tissue samples collected during surgical procedures, as compared to hypogonadal untreated subjects and eugonadal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Age between 25 and 65 years
* Obese men, candidate to a bariatric surgery (body mass index (BMI) is ≥40 kg/m2, or if their BMI is >35 kg/m2 and they suffer from other life-threatening co-morbidities such as Type 2 Diabetes Mellitus, hypertension and cardiovascular disease)
* Men with LUTS defined by: IPSS ≥ 8.
* Evidence of a personally signed and dated informed consent

Exclusion Criteria:

* Bladder failure or Neurogenic bladder
* LUT disease (Urethral stenosis, diverticula)
* LUT surgery (Prostatectomy, bladder neck surgery, TURP)
* Severe systemic disease
* Previous or concomitant neoplasm
* Unable to consistently and accurately complete the protocol
* Abuse alcohol or drugs
* Psychiatric disease

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male adults subjects suffering from severe obesity in a waiting list for bariatric surgery for weight loss will be considered eligible.
  The diagnosis of hypogonadism will be defined by levels of total testosterone <12nmol / l or free testosterone <225 pmol / L (calculated according to the formula of Vermeulen).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
IPSS score (LUTS) improvement | 1 yr after surgery
  For each patient the presence of an improvement of LUTS, assessed by IPSS score, will be evaluated by calculating the difference between the scores of the IPSS questionnaire administered at V1 compared to that administered to V0, V2 as compared to V1, or V3 as compared to V2. The mean of this change will be then compared between different groups (eugonadal; untreated hypogonadal; treated hypogonadal)

SECONDARY OUTCOMES:
Presence of Metabolic Syndrome | 1 yr after surgery
  The diagnosis of MetS parameters will be re-evaluated to confirm the presence or absence (waist circumference, dyslipidemia, blood pressure, fasting plasma glucose)
Volumetric change of the prostate | 1 yr after surgery
Change in the number of prostatic macrocalcifications | 1 yr after surgery
Change in the peak of arterial velocity at the colour-doppler ultrasound of the prostate | 1 yr after surgery
Improvement of sexual function | 1 yr after surgery
  Improvement of sexual function will be assessed by evaluating differences in the score obtained at the IIEF-5 (International Index of Erectile Function), a questionnaire which assesses erectile function by 5 questions with a score from 0 to 5, by giving 5 to the best erectile function. Scores range from 1 to 25, and a cut-off of 21 defines erectile dysfunction (score <21).
Improvement of symptoms of hypogonadism | 1 yr after surgery
  Improvement of sexual function will be assessed by evaluating differences in the score obtained at the AMS (Aging Male's symptoms). This questionnaire consists of 17 questions which investigate the disturbances of the psychological, somatic and sexual domain; for each question the patient gives a numerical answer ranging from 1 (no symptoms) to 5 (very severe symptoms). The assessment of symptoms is obtained from the numerical sum of 17 responses. The symptoms are classified as: • absent: score 17 to 26; • mild: score 27 to 36; • moderate: score 37 to 49; • severe: score ≥ 50.
Preadipocyte dysfunction assessed in preadipocyte isolated from visceral adipose tissue obtained during bariatric surgery | 1 yr after surgery
Variations in histomorphometric and molecular parameters of hepatic tissue obtained during bariatric surgery | 1 yr after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maggi, Principal Investigator — University of Florence
Locations (1):
- Ambulatori Medicina della Sessualità e Andrologia, Florence, Italy

REFERENCES:
- [Background] Lotti F, Corona G, Colpi GM, Filimberti E, Degli Innocenti S, Mancini M, Baldi E, Noci I, Forti G, Adorini L, Maggi M. Elevated body mass index correlates with higher seminal plasma interleukin 8 levels and ultrasonographic abnormalities of the prostate in men attending an andrology clinic for infertility. J Endocrinol Invest. 2011 Nov;34(10):e336-42. doi: 10.3275/7855. Epub 2011 Jul 7. PMID 21738005
- [Background] Filippi S, Vignozzi L, Morelli A, Chavalmane AK, Sarchielli E, Fibbi B, Saad F, Sandner P, Ruggiano P, Vannelli GB, Mannucci E, Maggi M. Testosterone partially ameliorates metabolic profile and erectile responsiveness to PDE5 inhibitors in an animal model of male metabolic syndrome. J Sex Med. 2009 Dec;6(12):3274-88. doi: 10.1111/j.1743-6109.2009.01467.x. Epub 2009 Sep 1. PMID 19732305
- [Background] Vignozzi L, Morelli A, Sarchielli E, Comeglio P, Filippi S, Cellai I, Maneschi E, Serni S, Gacci M, Carini M, Piccinni MP, Saad F, Adorini L, Vannelli GB, Maggi M. Testosterone protects from metabolic syndrome-associated prostate inflammation: an experimental study in rabbit. J Endocrinol. 2012 Jan;212(1):71-84. doi: 10.1530/JOE-11-0289. Epub 2011 Oct 18. PMID 22010203
- [Derived] Maseroli E, Comeglio P, Corno C, Cellai I, Filippi S, Mello T, Galli A, Rapizzi E, Presenti L, Truglia MC, Lotti F, Facchiano E, Beltrame B, Lucchese M, Saad F, Rastrelli G, Maggi M, Vignozzi L. Testosterone treatment is associated with reduced adipose tissue dysfunction and nonalcoholic fatty liver disease in obese hypogonadal men. J Endocrinol Invest. 2021 Apr;44(4):819-842. doi: 10.1007/s40618-020-01381-8. Epub 2020 Aug 8. PMID 32772323